CLINICAL TRIAL: NCT01415999
Title: Novel Imaging and Circulation Biomarkers for Comprehensive Evaluation of Cardiovascular Function in Adult Survivors of Childhood Malignancies
Brief Title: Cardiovascular Function in Adult Survivors of Childhood Malignancies
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Yiu-fai Cheung, Professor, The University of Hong Kong
Other Study IDs: UW 11-289
Record Dates: First submitted 2011-08-10; First posted 2011-08-12 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Childhood Cancers
Keywords: anthracycline; cardiac function; echocardiography; biomarkers

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — plasma, serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- patient: adult survivors of childhood malignancies
- control: healthy age-matched individuals

SUMMARY:
Anthracyclines have been used commonly to treat children with solid tumours and haematological malignancies and have led to their increased survival. Nonetheless, anthracycline has the side effect of cardiotoxicity. The purpose of this study is to assess the impact of anthracycline therapy on heart deformation and fibrosis, heart-vessel interaction, usefulness of circulating biomarkers in the assessment of heart function and potential genetic predisposition to heart failure in adult survivors of childhood cancers.

DETAILED DESCRIPTION:
Incorporation of anthracyclines into chemotherapy protocols has improved the survival of children with solid tumours and haematological malignancies. Nonetheless, longitudinal studies have implicated the absence of a safe anthracycline dose that is free of cardiotoxicity. Substantial risk for cardiovascular disease has been shown recently in large cohorts of adult survivors of childhood and adolescent survivors. Serial monitoring of cardiac function is hence of paramount importance in childhood cancer survivors for early detection of myocardial damage and timely institution of interventions. The optimal monitoring of cardiac function in the long term in these at-risk patients remains to be established. Novel noninvasive imaging modalities including echocardiography and cardiac magnetic resonance allow interrogation of myocardial deformation and fibrosis, while circulating biomarkers are increasingly used to monitor the cardiac status in heart failure patients. Additionally, genetics of heart failure are increasingly unveiled.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 to 35 years old
* history of acute leukaemia diagnosed before 18 years old
* completion of cancer directed therapy for at least 5 years.

Exclusion Criteria:

* history of congenital heart disease
* presence of syndromal disorder such as Down syndrome, neurofibromatosis, etc,
* hypothyroidism not on replacement therapy
* claustrophobia or other reasons rendering MRI assessment not feasible.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients will be recruited from the 5 public hospitals in Hong Kong (Prince of Wales Hospital, Princess Margaret Hospital, Queen Elizabeth Hospital, Queen Mary Hospital, and Tuen Mun Hospital) that treat the vast majority of childhood cancers, with the number of patients recruited from each hospital proportional to the respective new case-loads in the past 10 years.
Sampling Method: Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yiu-fai Cheung, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong, China